CLINICAL TRIAL: NCT06987942
Title: A Randomized, Controlled, Phase Ⅳ Clinical Trial to Evaluate the Immunogenicity and Safety of Live Attenuated Varicella Vaccine Administered Concomitantly With Trivalent Inactivated Influenza Vaccine (Split Virion) in Children Aged 7-12 Years
Brief Title: Simultaneous Administration Study of Varicella Attenuated Live Vaccine and Trivalent Inactivated Influenza Vaccine (Split Virion)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-VAR-MA4004-JS-2
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Varicella; Influenza Vaccine
MeSH Terms: conditions — Chickenpox; Influenza, Human | interventions — Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simultaneous vaccination group (Experimental): Participants received a single dose of varicella vaccine and TIV on Day 0.
  Interventions: Biological: Varicella vaccine+TIV
- Varicella vaccine separate group (Active Comparator): Participants received a single dose of varicella vaccine on Day 0.
  Interventions: Biological: Varicella vaccine
- TIV separate group (Active Comparator): Participants received a single dose of TIV on Day 0.
  Interventions: Biological: TIV

INTERVENTIONS:
Biological: Varicella vaccine+TIV — * Varicella vaccine: lyophilized powder, subcutaneous injection
  * TIV: Inactived, split virion, containing H1N1, H3N2 and BV strains.
  Arms: Simultaneous vaccination group
Biological: Varicella vaccine — lyophilized powder, subcutaneous
  Arms: Varicella vaccine separate group
Biological: TIV — Inactived, split virion, containing H1N1, H3N2 and BV strains.
  Arms: TIV separate group

SUMMARY:
The goal of this clinical trial is to evaluate the immunogenicity of simultaneous administration of varicella live attenuated vaccine (varicella vaccine hereafter) and trivalent inactivated influenza vaccine (TIV hereafter). It will also evaluate the safety of simultaneous administration of the two vaccines. The main questions it aims to answer are:

* If geometric mean titer (GMT) of varicella zoster vrius (VZV) antibody in the simultaneous administration group is non-inferior to that in the varicella vaccine separate group.
* If GMT of hemagglutination inhibition (HI hereafter) antibody in the simultaneous administration group is non-inferior to that in the TIV separate group.

Participants in the simultaneous administration group received a single dose of varicella vaccine and TIV simultaneously on day 0. Participants in the separate groups received a single dose of varicella vaccine or TIV on day 0, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 7-12 years;
* The subject or legal guardian can understand and sign the informed consent form (double signature is required for those over 8 years old);
* Participants and their legal guardians voluntarily participate in the study and are able to comply with all study procedures;
* Provide legal identity proof;

Exclusion Criteria:

* Vaccination history of varicella vaccine;
* Had received a single dose of influenza vaccine for 2024-2025 season;
* History of varicella;
* History of severe allergic reactions to vaccines (such as acute anaphylaxis, angioedema, dyspnea, etc.);
* Suffering from acute disease, severe chronic disease, acute exacerbation of chronic disease;
* With any confirmed or suspected immunodeficiency disease, immunocompromised or receiving immunosuppressive therapy (including systemic steroid therapy);
* With a history of congenital immune diseases or close contact with family members with a history of congenital immune diseases;
* With encephalopathy, uncontrolled epilepsy, other progressive neurological disorders, history of Guillain-Barre syndrome;
* Body temperature >37℃ at the time of vaccination;
* Receipt of blood products within 3 months before receiving investigational vaccine;
* Receipt of another study drug within 30 days before receipt of the investigational vaccine;
* Receipt of live attenuated vaccine within 28 days before receipt of investigational vaccine;
* Receipt of subunit or inactivated vaccine within 7 days before receipt of investigational vaccine;
* Participated in other clinical trials before enrollment and were enrolled in another clinical trial during the follow-up period or planned to participate in another clinical trial within 3 months;
* The participant had any other factors that were ineligible for vaccination by in the investigator's judgment.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 899 (Actual)
Dates: Start 2024-09-21 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
GMT of VZV antibody | Day 30 after the vaccination
  GMT of VZV antibody on Day 30 after the vaccination.
GMT of HI antibody | Day 30 after vaccination
  GMT of HI antibody on Day 30 after vaccination.

SECONDARY OUTCOMES:
Geometric mean increase (GMI) of VZV antibody | Day 30 after the vaccination
  GMI of VZV antibody on Day 30 after the vaccination.
Seroconversion rate of VZV antibody | Day 30 after the vaccination
  Seroconversion rate of VZV antibody on Day 30 after the vaccination.
Seropositive rate of VZV antibody | Day 30 after the vaccination
  Seropositive rate of VZV antibody on Day 30 after the vaccination.
GMI of HI antibody | Day 30 after the vaccination
  GMI of HI antibody on Day 30 after the vaccination.
Seroconversion rate of HI antibody | Day 30 after the vaccination
  Seroconversion rate of HI antibody on Day 30 after the vaccination.
Seroprotection rate of HI antibody | Day 30 after the vaccination
  Seroprotection rate of HI antibody on Day 30 after the vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Disease control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No